CLINICAL TRIAL: NCT01669070
Title: An Open Label, Part-randomised, Four-way Crossover, Single and Repeat Dose Study to Determine the Dose Proportionality and Absolute Bioavailability of Fluticasone Furoate (FF) When Administered as FF Inhalation Powder From the Novel Dry Powder Inhaler in Healthy Subjects
Brief Title: A Four-way Crossover, Single and Repeat Dose Study to Determine the Dose Proportionality and Absolute Bioavailability of Fluticasone Furoate Inhalation Powder Administered by Novel Dry Powder Inhaler (NDPI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115441
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: bioavailability; Fluticasone Furoate; pharmacokinetics; dose proportionality
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FF 50 mcg powder inhalation (Experimental): Each subject will receive a single dose of 300 mcg FF (6 inhalations of 50 mcg FF) on Day 1 of the respective period per randomization sequence, followed by 50 mcg FF once daily for 7 days, on Days 3-9 inclusive, administered from the NDPI.
  Interventions: Drug: FF, 50 mcg
- FF 100 mcg powder inhalation (Experimental): Each subject will receive a single dose of 600 mcg FF (6 inhalations of 100 mcg FF) on Day 1 of the respective period per randomization sequence, followed by 100 mcg FF once daily for 7 days, on Days 3-9 inclusive, administered from the NDPI.
  Interventions: Drug: FF, 100 mcg
- FF 200 mcg powder inhalation (Experimental): Each subject will receive a single dose of 1200 mcg FF (6 inhalations of 200 mcg FF) on Day 1 of the respective period per randomization sequence, followed by 200 mcg FF once daily for 7 days, on Days 3-9 inclusive, administered from the NDPI.
  Interventions: Drug: FF, 200 mcg
- FF 250 mcg IV (Experimental): Each subject will receive a single dose of 250 mcg FF, administered as an IV infusion over 20 minutes on Day 1 of the respective period per randomization sequence.
  Interventions: Drug: FF, 250 mcg

INTERVENTIONS:
Drug: FF, 50 mcg — Novel dry powder inhaler
  Arms: FF 50 mcg powder inhalation
Drug: FF, 100 mcg — Novel dry powder inhaler
  Arms: FF 100 mcg powder inhalation
Drug: FF, 200 mcg — Novel dry powder inhaler
  Arms: FF 200 mcg powder inhalation
Drug: FF, 250 mcg — Intravenous
  Arms: FF 250 mcg IV

SUMMARY:
The purpose of this study is to demonstrate dose proportionality of the FF (50 microgram (mcg), 100 mcg or 200 mcg), when administered as a single and repeat dose from the NDPI containing FF formulated with lactose. In addition, the aim of this study is to determine the absolute bioavailability of the FF single strip product using the high strength product administered as a single dose with multiple inhalations and using 250 mcg intravenous (IV) FF.

This is a, part-randomized, open-label, 4 way crossover study (4 periods) in healthy adult subjects. During each period, subjects will receive FF in the morning and serial pharmacokinetic (PK) sampling (for up to 10 days for the inhaled treatment and up to 3 days for the IV treatment) and safety assessments will be performed. Each period will be separated by a washout period of at least 7 days and a follow-up telephone call will occur 7 -14 days after the last dose of study drug. The total duration of the study will be approximately 13-14 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18 and 65 years of age and body mass index (BMI) within the range 18.5 to 29.0 kilogram/meter squared.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) and bilirubin < or =1.5x upper limit of normal (ULN).
* Female subjects of child bearing potential are eligible to enter if they are not pregnant and willing to use protocol-specified methods of contraception to prevent pregnancy during the study.
* Average QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 millisecond.
* Forced Expiratory Volume in 1 Second (FEV1) > or = 85% predicted at screening.
* Current non-smokers
* Able to satisfactorily use the NDPI.

Exclusion Criteria:

* Subjects must not have a systolic blood pressure above 145 milimeter(mm) of mercury(Hg) or a diastolic pressure above 85 mmHg at the screening visit.
* History of breathing problems in adult life confirmed by normal lung function parameters (≥85% predicted).
* Donation of more than 500 mL blood within a 56 day period.
* Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* The subject treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* The subject has a positive: drug/alcohol, Hepatitis, HIV screen.
* Abuse of alcohol.
* Subject having positive cotinine and urine alcohol test.
* Participated in >3 clinical trials in the previous 10 months (if male), or >2 clinical trials in the previous 10 months (if female), or the subject has participated in a study (including follow up) within 60 days prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Taken systemic, oral or depot corticosteroids less than 12 weeks or inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* Use of prescription or non-prescription drugs.
* History of severe milk protein allergy, sensitivity to any of the study medications, including immediate or delayed hypersensitivity to any intranasal, inhaled or systemic corticosteroid therapy.
* Pregnant or lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2012-11-16 (Actual)

PRIMARY OUTCOMES:
FF pharmacokinetics; parameters: (AUC(0-infinity)) , (AUC(0-24)) and (Cmax) | 54 days
  FF pharmacokinetics; area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC (0-infinity)), area under the concentration-time curve from zero (pre-dose) to 24 h (AUC (0-24)) and maximum observed concentration (Cmax). Blood samples for PK analysis of FF will be collected and analysis will be performed. Concentrations of FF will be determined in plasma samples using the currently approved analytical methodology.

SECONDARY OUTCOMES:
Plasma FF PK parameters: t1/2, tmax, MRT for all treatments | 54 days
  Following plasma FF PK parameters will be evaluated: terminal phase half life (t1/2), time of occurrence of Cmax (tmax), mean residence time (MRT) for all treatments Blood samples for PK analysis of FF will be collected and analysis will be performed. Concentrations of FF will be determined in plasma samples using the currently approved analytical methodology.
Plasma FF PK parameters: V and CL for IV treatment | 3 days (Study Day 52 to Study Day 54)
  Following plasma FF PK parameters will be evaluated: volume of distribution (V) and plasma clearance (CL) for intravenous administration Blood samples for PK analysis of FF will be collected and analysis will be performed. Concentrations of FF will be determined in plasma samples using the currently approved analytical methodology.
Mean absorption time (MAT) for inhaled treatments | 44 days
  Blood samples for PK analysis of FF will be collected and analysis will be performed. Concentrations of FF will be determined in plasma samples using the currently approved analytical methodology.
Safety of FF | 68 days
  To assess the safety and tolerability of FF administered as single and repeat dose adverse events will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115441 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115441?search=study&search_terms=115441#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115441 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register